CLINICAL TRIAL: NCT05822219
Title: Leveraging Community-Academic Partnerships and Social Networks to Disseminate Vaccine-Related Information and Increase Vaccine Uptake Among Black Individuals With Rheumatic Diseases.
Brief Title: Vaccine Hesitancy in Black/African Americans With Rheumatic Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Rosalind Ramsey-Goldman, Principal Investigator - Chicago, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ACTIVATE
Record Dates: First submitted 2023-03-20; First posted 2023-04-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Rheumatic Diseases; COVID-19 Vaccine; COVID-19; SLE
Keywords: Social network; Community based intervention; Vaccine uptake; Popular Opinion Leaders
MeSH Terms: conditions — Rheumatic Diseases; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Intervention Model Description: Two different group training arms related to COVID-19 vaccine uptake
Masking Description: Participants are unblinded but study has non-disclosure component of keeping the difference between the two training arms as non-disclosed until the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COVID-19 vaccine and booster training (Active Comparator): Group training involving COVID-19 vaccine and booster information, including background, development, and myths.
  Interventions: Behavioral: COVID-19 vaccine and booster training, and importance
- COVID-19 vaccine and booster training with extra undisclosed component (Experimental): Group training involving COVID-19 vaccine and booster information, including background, development, and myths. Contains extra training component that is undisclosed until the end of the study so as not to introduce bias.
  Interventions: Behavioral: COVID-19 vaccine and booster training, and importance

INTERVENTIONS:
Behavioral: COVID-19 vaccine and booster training, and importance — COVID-19 vaccine and booster information training

SUMMARY:
To establish the efficacy of a community-based POL (Popular Opinion Leader) intervention with two different trainings designed to increase COVID-19 vaccine and booster uptake and reduce hesitancy among social networks of Black individuals with rheumatic conditions. The investigators will also determine the structure and composition of the personal and outreach social networks of POLs.

DETAILED DESCRIPTION:
Through community-academic partnerships in Boston and Chicago, investigators will recruit and randomly assign POLs who identify as Black with rheumatic conditions to two training arms in each city. Arms 1 and 2 will receive the same core curriculum addressing COVID-19 vaccine hesitancy, safety and efficacy. POLs will work in their communities to distributed information they learned in the trainings to members of their social network. The investigators will gather information about these social networks, assessing for differences in characteristics such as size, location, and who is in it (percentage of family, percentage Black, percentage with rheumatic conditions).

ELIGIBILITY:
Inclusion Criteria:

POLs:

18-85 years old; All genders; English-speaking; Self-identify as Black and/or African descent; Received ≥1 dose of a COVID-19 vaccine after 8.31.2022 (bivalent booster or updated COVID-19 vaccine [2023-2024] formula)

Social network members:

At least 18 years of age; All genders; English-speaking or Haitian Creole or Spanish-speaking if the POL also speaks Haitian Creole or Spanish; Not have received the updated COVID-19 vaccine 2023-2024 formula; Recent (within 3 months) COVID-19 infection and either undecided or no intention of receiving the vaccine.

Exclusion Criteria:

Both POLs and social network members:

Under 18 years of age Pregnant women Institutionalized or incarcerated Those who are up to date on COVID vaccinations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Receipt of >1 COVID-19 vaccine or booster dose | 6 months
  This will be measured as documentation of receipt of >1 additional COVID-19 vaccine or booster dose above network members' baseline number of doses, scored yes or no.

SECONDARY OUTCOMES:
Change in COVID-19 vaccine hesitancy | 6 months
  This will be measured as the network members' absolute change in vaccine hesitancy scale score comparing 6 months to baseline between the two study arms, using the validated 10-item Likert Vaccine Hesitancy Scale, score range 10-50.
Structure and composition of the Popular Opinion Leader outreach networks. | 6 months
  A mixed methods social network assessment tool will be used to compare the structures and compositions of the outreach social networks of the Popular Opinion Leaders between the two intervention arms. This is not scored but rather used to create social network map and to understand characteristics of social networks.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, MD, DrPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The final data sets from this project will include participant reported survey outcomes and will be de-identified in accordance with HIPAA guidelines. Several methods of resource sharing will be employed by this project including:1)Publishing of results in scientific journals and presentation at professional meetings 2)Replies to requests from individuals for data, and sent via secure methods such as password protected files 3)Posting of POL training curriculum after all data are collected on Dr. Ramsey-Goldman's (MPI) NU webpage 4)Posting study-specific adaptations made to social network survey on website of Dr. Dhand (Co-Investigator).
Supporting Information: Study Protocol
Time Frame: Resource sharing will be made available in a timely manner and no later than 12 months after the publication of the main findings from the final data set.
Access Criteria: Any investigator who wishes to obtain data from this Project will do so with a Resource Sharing Agreement that provides for 1) a commitment to using the resources only for research purposes and not to identify an individual participant.2) a commitment to securing resources using appropriate computer technology.3) a commitment to destroy or return the resources after analyses are completed.4) cover the cost of preparing data including programming time and other tasks required to transfer the dataset.

REFERENCES:
- [Derived] Sirek G, Erickson D, Muhammad LN, Losina E, Chandler MT, Son MB, Crespo-Bosque M, York M, Jean-Jacques M, Milaeger H, Pillai N, Roberson T, Chung A, Shramuk M, Osaghae E, Williams J, Ojikutu BO, Dhand A, Ramsey-Goldman R, Feldman CH. Community-engaged randomised controlled trial to disseminate COVID-19 vaccine-related information and increase uptake among Black individuals in two US cities with rheumatic conditions. BMJ Open. 2024 Aug 24;14(8):e087918. doi: 10.1136/bmjopen-2024-087918. PMID 39181556
- [Derived] Sirek G, Ulysse S, Jacques Toussaint M, Nosamiefan C, Desrosiers L, Chandler M, Ramsey-Goldman R, Fleurissaint DJ, Feldman CH. A community-engaged approach to translate a Vaccine Hesitancy Scale into Haitian Creole. Vaccine. 2024 Apr 2;42(9):2127-2134. doi: 10.1016/j.vaccine.2024.02.079. Epub 2024 Mar 7. PMID 38458871